CLINICAL TRIAL: NCT06931262
Title: Expanded Access Treatment Protocol With Dichloroacetate Sodium for Patients With Pyruvate Dehydrogenase Complex Deficiency
Brief Title: Expanded Access Treatment Protocol With DCA for Patients With PDCD
Status: Available | Type: Expanded Access
Sponsor: Saol Therapeutics Inc (Industry)
Collaborators: AnovoRx (Unknown)
Responsible Party: Sponsor
Other Study IDs: SL 1009 EA-01
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency
Keywords: PDCD
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease | interventions — Dichloroacetic Acid

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Dichloroacetate (DCA) — Study medication DCA is an oral solution mixed with an artificial sweetener containing aspartame and strawberry extract (50mg/mL) Participants will be genotyped to determine GSTZ1 (glutathione S-transferase Zeta-1) haplotype status, which will stratify this group into 1 of 2 dose regimens: EGT carriers will receive 12 mg/kg/12hr DCA. EGT non-carriers will receive 6 mg/kg/12 hr DCA.

SUMMARY:
Expanded Access (EA) will provide a transition to continue therapy for those patients who are currently in the open label extension of the Phase III study, SL 1009-01, while also allowing new patients diagnosed with PDCD who meet the eligibility criteria to also have access to therapy that would be otherwise unavailable.

DETAILED DESCRIPTION:
Expanded Access (EA) will provide a transition to continue therapy for those patients who are currently in the open label extension of the Phase III study, SL 1009-01, while also allowing new patients diagnosed with PDCD who meet the eligibility criteria to also have access to therapy that would be otherwise unavailable. The Expanded Access program (EAP) will also allow the sponsor to extend the collection of long term safety data for the current open label patients, while also expanding to an additional population of patients beyond those currently in the SL 1009-01 study.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 0 through adulthood
2. Presence of characteristic clinical or metabolic features of PDCD and
3. Presence of a known pathogenic mutation of a gene that is specifically associated with PDC (PDHA1, PDHB, DLAT, PDHX, DLD).
4. Females of reproductive age must be willing to use an effective method of barrier contraception for the duration of the study.-

Exclusion Criteria:

1. A genetic mitochondrial disease other than those stipulated under inclusion criteria
2. Primary, defined organic acidurias other than lactic acidosis (e.g., propionic aciduria)
3. Primary disorders of amino acid metabolism
4. Primary disorders of fatty acid oxidation
5. Secondary lactic acidosis due to impaired oxygenation or circulation (e.g., due to severe cardiomyopathy or congenital heart defects)
6. Malabsorption syndromes associated with D-lactic acidosis
7. Renal insufficiency, defined as 1) a requirement for chronic dialysis or 2) serum creatinine ≥ 1.2 mg/dl or creatinine clearance <60 ml/min
8. Primary hepatic disease unrelated to PDCD
9. Pregnancy or breast feeding -

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Diorgu, M.D., Study Chair — Saol Therapeutics Inc